CLINICAL TRIAL: NCT03904407
Title: Optimizing Overactive Bladder Treatment: A Randomized Trial Investigating the Influence of Probiotic Therapy on the Urinary Microbiome and Response to Anticholinergic or Beta-3 Agonist Therapy
Brief Title: Optimizing Overactive Bladder Treatment
Acronym: OPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Society of Urodynamics, Female Pelvic Medicine & Urogenital Reconstruction (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-0030
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; probiotic; anticholinergic; beta-3 agonist
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Sugars

STUDY DESIGN:
Intervention Model Description: Randomized double blind placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Probiotic study drug and identical appearing placebo tablet
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Lactobacillus probiotic capsules in addition to a routine-care prescribed anticholinergic or beta-3 agonist medication for 4 weeks.
  Interventions: Other: Lactobacillus Probiotic Capsule
- Placebo (Placebo Comparator): Matching Lactobacillus probiotic placebo capsules in addition to a routine-care prescribed anticholinergic or beta-3 agonist medication for 4 weeks.
  Interventions: Other: Matching Lactobacillus Probiotic Placebo Capsule

INTERVENTIONS:
Other: Lactobacillus Probiotic Capsule — One over-the-counter, probiotic capsule taken by mouth once daily for 4 weeks. Each capsule contains 10 billion cells comprised of:
  * Lactobacillus crispatus LbV 88
  * Lactobacillus jensenii LbV 116
  * Lactobacillus gasseri LbV 150N
  * Lactobacillus rhamnosus LbV 96
  Other Names: Jarro-Dophilus Women
  Arms: Probiotic
Other: Matching Lactobacillus Probiotic Placebo Capsule — Lactobacillus Probiotic placebo capsules identical in appearance taken by mouth once daily for 4 weeks
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Purpose: This is a pilot randomized double-blind placebo controlled trial of anticholinergic or beta-3 agonist medication with or without concomitant probiotic therapy in women initiating medication therapy for overactive bladder (OAB). The aims of this study are to:

1. Explore how concomitant probiotic therapy influences response to medication for OAB in a randomized controlled trial
2. Investigate whether 4 weeks of probiotic therapy alters the urinary microbiome
3. Assess for predictors of response to therapy

Participants: Women 18 years of age or older presenting to the Division of Urogynecology and Reconstructive Pelvic Surgery clinic with OAB/UUI or UUI-predominant mixed incontinence who desire nonsurgical therapy will be eligible for participation.

Procedures (methods): The study will be conducted over a two-year time frame and the primary outcome will be subjective improvement in symptoms as assessed by the Patient Global Impression of Improvement (PGI-I) validated questionnaire at 4 weeks after initiating anticholinergic or beta-3 agonist medication and study drug. The study aims to recruit up to 140 participants randomized in a 1:1 ratio to either concomitant probiotic or placebo medication.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a highly prevalent condition that negatively impacts the lives of millions of adults in the United States. Anticholinergic and beta-3 agonist medications are commonly used to treat OAB but compliance is low due to variable efficacy and bothersome side effects. The existence of a urinary microbiome was recently discovered and early investigations have revealed that lower Lactobacillus load is correlated with the presence of OAB symptoms and a poorer response to anticholinergic therapy.

This proposed pilot study is a randomized double-blind placebo-controlled trial (RCT) of concomitant probiotic therapy in women initiating medication therapy for OAB to explore how probiotics influence response to anticholinergic and beta-3 agonist medications, investigate whether probiotic therapy alters the urinary microbiome, and assess for predictors of response to therapy.

Primary Aim: To explore how concomitant probiotic therapy influences response to medication for OAB in a RCT

Secondary Aims:

1. To investigate whether 4 weeks of probiotic therapy alters the urinary microbiome.
2. To assess for predictors of response to therapy

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18 years
* English-speaking
* OAB/UUI or urge-predominant mixed incontinence per the Medical Epidemiologic and Social Aspects of Aging (MESA) questionnaire

Exclusion Criteria:

* Neurogenic bladder or urinary retention (postvoid residual (PVR) >150 mL)
* Probiotic use within the past 4 weeks
* Inflammatory bowel disease or history of bariatric surgery
* Pelvic organ prolapse past the hymen
* Current symptomatic UTI or systemic antibiotic exposure within 4 weeks
* Current treatment for recurrent UTI or history of recurrent UTI in the last 6 months
* Immunosuppressive therapy (i.e., prednisone or chemotherapy)
* Contraindication to anticholinergic or beta-3 agonist medication (including pregnancy)
* Prior neuromodulation therapy for OAB
* Inability or unwillingness to comply with study protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Success Based on the PGI-I Validated Questionnaire Response | 4 weeks
  Treatment success at 4 weeks after initiation of anticholinergic of beta-3 agonist therapy. Treatment success will be defined as a response of "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I), which is a single item questionnaire that asks respondents to rate their improvement after undergoing treatment on a 7-point Likert scale ranging from "very much worse" to "very much better." Statistical analysis will be by intention-to-treat for the primary outcome. A chi-square test will be utilized to determine if there is a statistically significant difference between the two cohorts and sensitivity analyses will be performed using logistic regression analysis.

SECONDARY OUTCOMES:
Change in participant's urinary microbiome from baseline to week 4 | Baseline, Week 4
  Each participants' urinary microbiome composition will be analyzed at baseline and at week 4 to determine changes in the microbiome that occur over the study period. The correlation between changes in the urinary microbiome over 4 weeks and study drug allocation (probiotic vs placebo) will be assessed via Chi-square testing.
Urinary microbiome Lactobacillus correlation with treatment success as defined by PGI-I Validated Questionnaire Response | 4 weeks
  The correlation between the presence of Lactobacillus in the urine at baseline and treatment success at week 4 will be analyzed via Chi-Square testing to assess for predictors of response to therapy in women (i.e. treatment success or lack of treatment success based on the primary outcome definition of treatment success as above).
OAB-Q SF Change Score | Baseline, Week 4
  Individual participant change score on the Overactive Bladder Questionnaire short-form (OAB-q SF) will be compared between the two cohorts by student's t-test. The OAB-q SF is utilized to assess the impact of OAB symptoms on the patient's life, and has been shown to be responsive to reductions in urinary urgency, frequency and incontinence during anticholinergic therapy. The OAB-q SF questionnaire consists of 19 items divided into a 6-item symptom severity (SS) scale and a 13-item health-related quality of life (HRQL) scale, with both scales ranging from 0 to 100. For the OAB-q SS scale a higher score indicates worse symptom severity while for the OAB-q HRQL scale a higher score indicates better quality of life.
TQSM-II Validated Questionnaire Score | Week 4 Visit
  Treatment Satisfaction Questionnaire for Medication version 2 (TQSM-II) score, the TQSM-II is comprised of 12 questions assessing treatment satisfaction with medication intended for use with a wide variety of medications and illness conditions that specifically assesses the three most common dimensions on which patients evaluate their medication: effectiveness, side effects of use, and convenience of use. TSQM Scale scores range from 0 to 100 with a higher score indicating better satisfaction with treatment. The TQSM-II score at the week 4 visit will be compared between the two cohorts by student's t-test.
Correlation between race/ethnicity and treatment success as Defined by PGI-I Validated Questionnaire Response | Week 4 Visit
  Treatment success will be defined as a response of "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I), which is a single item questionnaire that asks respondents to rate their improvement after undergoing treatment on a 7-point Likert scale ranging from "very much worse" to "very much better." The correlation between race/ethnicity and treatment response will be analyzed using chi-square or fisher's exact test.
Correlation between OAB medication dose and Lactobacillus Load in the Urinary Microbiome | Week 4
  The correlation between the presence of Lactobacillus in the urinary microbiome and dose of OAB medication at 4 weeks (i.e. low dose vs high dose) will be analyzed via Chi-square or fishers exact test.

OTHER OUTCOMES:
Per Protocol Analysis of Treatment Success as Defined by PGI-I Validated Questionnaire Response | Week 4
  Treatment success will be defined as a response of "very much better" or "much better" on the Patient Global Impression of Improvement (PGI-I), which is a single item questionnaire that asks respondents to rate their improvement after undergoing treatment on a 7-point Likert scale ranging from "very much worse" to "very much better." A per protocol analysis of treatment success at 4 weeks (the primary outcome) will also be performed using a chi-square test to determine if there is a statistically significant difference between the two cohorts in treatment success and sensitivity analyses may be performed using logistic regression analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Dieter, MD, Principal Investigator — The University of North Carolina at Chapel Hill School of Medicine
Locations (2):
- United States (2):
  - UNC Hillsborough Medical Office Building, Hillsborough, North Carolina
  - UNC Urogynecology and Reconstructive Pelvic Surgery, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared until 24 months following publication of the first manuscript from this study provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: Until 24 months following publication of the first manuscript from this study.
Access Criteria: The investigator who proposes to use the data has to have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.